CLINICAL TRIAL: NCT03578055
Title: Prospective Study for the Effects of Biphenyl Dimethyl Dicarboxylate and Ursodeoxycolic Acid Therapy on Liver Function and Quality of Life After Laparoscopic Cholecystectomy
Brief Title: BDD With UDCA Therapy After Laparoscopic Cholecystectomy
Acronym: BULQ-LC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Huisong Lee, Assistant Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BULQ-LC trial
Record Dates: First submitted 2018-06-25; First posted 2018-07-05 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Cholecystitis, Acute; Cholecystitis, Chronic
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis; Bronchiolitis Obliterans Syndrome | interventions — 7,7'-dimethoxy-(4,4'-bi-1,3-benzodioxole)-5,5'-dicarboxylic acid dimethyl ester; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BDD with UDCA (Active Comparator): Postoperative BDD with UDCA treatment
  Interventions: Drug: BDD with UDCA
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BDD with UDCA — Dosage: Udex 1 capsule, 3 times daily Time of administration: 30 minutes after meal Duration of administration: From the day before surgery to 4 weeks after surgery
  Other Names: UDEX
  Arms: BDD with UDCA
Drug: Placebo — Dosage: 1 capsule of placebo, 3 times daily Time of administration: 30 minutes after meal Duration of administration: From the day before surgery to 4 weeks after surgery
  Other Names: No UDEX
  Arms: Placebo

SUMMARY:
Prospective Study for the Effects of Biphenyl Dimethyl Dicarboxylate and Ursodeoxycolic Acid Therapy on Liver Function and Quality of Life After Laparoscopic Cholecystectomy

Primary endpoint: peak level of postoperative AST (aspartate transaminase) and postoperative ALT (alanine tansaminase)

Secondary endpoint: postoperative GIQLI (Gastrointestinal Quality of Life index) score

DETAILED DESCRIPTION:
Because the gallbladder is adjacent to the liver, liver enzymes are often elevated when cholecystitis occurs. BDD and UDCA drugs are known to be effective in preserving liver function. The use of BDD and UDCA drugs in patients with cholecystitis is expected to inhibit elevated liver enzyme levels and to maintain liver function. The aim of this study is to analyze the effects of BDD and UDCA medication on postoperative changes in hepatic enzyme levels and quality of life in patients LFT elevated cholecystitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery due to chronic cholecystitis and acute cholecystitis

Exclusion Criteria:

* Failure to obtain consent
* Under 19 years
* If you have intellectual ability to understand this study
* When performing cholecystectomy with other operations
* Total bilirubin levels> 2 mg / dl
* If you are enrolled in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum Aspartate Aminotransferase | Postoperative 30 days
  Serum aspartate aminotransferase level (U/ml) (continuous variable)
Serum Alanine Aminotransferase | Postoperative 30 days
  Serum Alanine Aminotransferase level (U/ml) (continuous variable)

SECONDARY OUTCOMES:
GIQLI (Gastrointestinal Quality of Life Index) | Postoperative 30 days
  Score of Quastionare for postoperative quality of life by GIQLI (Range, 0 - 180)

CONTACTS AND LOCATIONS:
Overall Officials: Huisong Lee, M.D., Ph.D., Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No